CLINICAL TRIAL: NCT05456906
Title: Avoidable Hospitalizations/ Emergency Department Visits- Meta-synthesis of Qualitative Research
Brief Title: Avoidable Hospitalizations/ Emergency Department Visits- Systematic Review and Meta-synthesis of Qualitative Research
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University (Other)
Collaborators: The Ministry of Science and Technology (Unknown); National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Hsueh-Fen Chen, Associate Professor, Kaohsiung Medical University
Other Study IDs: 11; MOST110-2410-H-037-018-MY3 (Other Grant/Funding Number: Ministry of Science and Technology in Taiwan)
Record Dates: First submitted 2022-06-30; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Diabetes; Heart Failure; Chronic Obstructive Pulmonary Disease; Asthma; Hypertension; Urinary Tract Infections; Pneumonia, Bacterial
Keywords: Meta-analysis; Qualitative study; Systematic review; social determinants of health
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Hypertension; Urinary Tract Infections; Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No interventions

SUMMARY:
The aim of the study is to synthesize qualitative evidence related to preventable hospitalizations/ emergency department visits from the perspectives of patients, their families/caregivers, health care providers, and stakeholders, in the hope to identify generalizable conclusions about why social risk factors matter to preventable hospitalizations/ emergency department visits

DETAILED DESCRIPTION:
The present study is a qualitative systematic review and meta-synthesis study. The study primarily focused on the qualitative studies that collected and analyzed narratives from patients who experienced preventable hospitalizations. The information from their families, health care providers, and stakeholders in the qualitative studies are also included. The data collections from patients occurred during their hospital stay, emergency department stay, or after discharge to the community are included. Patients included all ages and gender, regardless of their race/ethnicity and countries.

The qualitative studies must be published in peer-reviewed journals, with language as english and no restriction on publication date or country of origin. Two authors (HC and HL) independently screened the title and reviewed abstracts, then full texts for eligibility. Thorugh synthesizing, the present study is expected to develop themes and sub-themes related to preventable hospitalizations/emergency department visits, in the hope to assist policymakers health care professionals, and stakeholders in properly addressing the underlying factors leading to preventable hospitalizations/emergency department visits .

ELIGIBILITY:
Patients were admitted to hospitals and/ or visited the emergency department due to preventable conditions, including diabetes acute complications, diabetes chronic complications, uncontrolled diabetes, low-extremity amputation due to diabetes, COPD, heart failure, hypertension, urinary tract infection, and pneumonia. Patients' families and their health care providers are also included.

exclusion criteria: patients with dementia, mental illness, or cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who experienced preventable hospitalizations and/ or emergency department visits, their families, and health care providers, with no restriction on publication date or country of origin, are included, regardless of their ages, gender, race/ethnicity, and country of birth.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
preventable hospitalizations and/or preventable emergency department visits | Patients were hospitalized or visited emergency department visits as the base line. The interviews were conducted during patient inpatient stay/ emergency department stay or after discharge to the community up to 3 years.
  patients who experienced hospitalizations and/ or emergency department visits due to any of the conditions: diabetes-related complication, heart failure, asthma, COPD, urinary tract infection, and bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh-Fen Chen, Ph.D., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
contact the corresponding author for reasonable reasons

REFERENCES:
- [Result] Granger BB, McBroom K, Bosworth HB, Hernandez A, Ekman I. The meanings associated with medicines in heart failure patients. Eur J Cardiovasc Nurs. 2013 Jun;12(3):276-83. doi: 10.1177/1474515112447734. Epub 2012 May 30. PMID 22653088
- [Result] James S, Annetts K, Frakking T, Broadbent M, Waugh J, Perry L, Lowe J, Clark S. Diabetic ketoacidosis presentations in a low socio-economic area: are services suitable? BMC Health Serv Res. 2021 Jul 10;21(1):682. doi: 10.1186/s12913-021-06715-7. PMID 34246266
- [Result] Longman JM, Rix E, Johnston JJ, Passey ME. Ambulatory care sensitive chronic conditions: what can we learn from patients about the role of primary health care in preventing admissions? Aust J Prim Health. 2018 Aug;24(4):304-310. doi: 10.1071/PY17191. Epub 2018 Aug 6. PMID 30078392
- [Result] Pasciak WE, Berg DN, Cherlin E, Fried T, Lipska KJ. Qualitative analysis of reasons for hospitalization for severe hypoglycemia among older adults with diabetes. BMC Geriatr. 2021 May 17;21(1):318. doi: 10.1186/s12877-021-02268-w. PMID 34001014
- [Result] Quensell ML, Taira DA, Seto TB, Braun KL, Sentell TL. "I Need my Own Place to get Better": Patient Perspectives on the Role of Housing in Potentially Preventable Hospitalizations. J Health Care Poor Underserved. 2017;28(2):784-797. doi: 10.1353/hpu.2017.0074. PMID 28529224
- [Result] Sentell TL, Seto TB, Young MM, Vawer M, Quensell ML, Braun KL, Taira DA. Pathways to potentially preventable hospitalizations for diabetes and heart failure: a qualitative analysis of patient perspectives. BMC Health Serv Res. 2016 Jul 26;16:300. doi: 10.1186/s12913-016-1511-6. PMID 27456233
- [Result] Shearer JE, Jenkins CH, Magwood GS, Pope CA. Contested Ownership of Disease and Ambulatory-Sensitive Emergency Department Visits for Type 2 Diabetes. Am J Med Sci. 2016 Apr;351(4):400-6. doi: 10.1016/j.amjms.2016.01.007. PMID 27079346
- [Result] van den Broek S, Heiwegen N, Verhofstad M, Akkermans R, van Westerop L, Schoon Y, Hesselink G. Preventable emergency admissions of older adults: an observational mixed-method study of rates, associative factors and underlying causes in two Dutch hospitals. BMJ Open. 2020 Nov 20;10(11):e040431. doi: 10.1136/bmjopen-2020-040431. PMID 33444202
- [Result] Manski-Nankervis JA, Furler J, Audehm R, Blackberry I, Young D. Potentially preventable hospitalisations: are they a useful marker of access to and experience of care in general practice among people with type 2 diabetes? Aust J Prim Health. 2015;21(2):214-20. doi: 10.1071/PY13112. PMID 24491142
- [Result] Ridge A, Peterson GM, Seidel BM, Anderson V, Nash R. Rural Patients' Perceptions of Their Potentially Preventable Hospitalisation: A Qualitative Study. J Patient Exp. 2022 Jan 4;9:23743735211069825. doi: 10.1177/23743735211069825. eCollection 2022. PMID 35005222
- [Result] McKenna G, Rogers A, Walker S, Pope C. The influence of personal communities in understanding avoidable emergency department attendance: qualitative study. BMC Health Serv Res. 2020 Sep 21;20(1):887. doi: 10.1186/s12913-020-05705-5. PMID 32958065
- [Result] Agarwal S, Banerjee J, Baker R, Conroy S, Hsu R, Rashid A, Camosso-Stefinovic J, Sinfield P, Habiba M. Potentially avoidable emergency department attendance: interview study of patients' reasons for attendance. Emerg Med J. 2012 Dec;29(12):e3. doi: 10.1136/emermed-2011-200585. Epub 2011 Dec 28. PMID 22205782
- [Derived] Chen HF, Lin HR. Social determinants of ambulatory care sensitive conditions: a qualitative meta-synthesis based on patient perspectives. Front Public Health. 2023 May 9;11:1147732. doi: 10.3389/fpubh.2023.1147732. eCollection 2023. PMID 37228726